CLINICAL TRIAL: NCT00295100
Title: Cancer Risk and Biomarkers of Tamoxifen Chemoprevention
Brief Title: Tamoxifen-MRI Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 278100; UPC 2100
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2007-06-21 (Estimated); Status verified 2007-06

CONDITIONS: Breast Cancer
Keywords: Tamoxifen; Prevention; Breast Cancer; MRI
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen

SUMMARY:
The project is a double blind, randomized, placebo-controlled phase II chemoprevention trial. Study participants will be randomly assigned to receive either tamoxifen or placebo for one year. Participants will subsequently be followed for one year off of medication. The primary objective is to evaluate the effectiveness of tamoxifen in reducing breast density by mammogram.

DETAILED DESCRIPTION:
The project is a double blind, randomized, placebo-controlled phase II chemoprevention trial.

The study outcomes will be biological markers, rather than cancer incidence or mortality. Eligible study subjects will be women, between the ages 25-45, whose calculated lifetime breast cancer risk is > 20% (25% by the Couch model).

Study participants will be randomly assigned to receive either tamoxifen or placebo for one year. Participants will subsequently be followed for one year off of medication.

The primary objective is to evaluate the effectiveness of tamoxifen in reducing breast density by mammogram. Mammographic density has been correlated with breast cancer risk and reduced breast density may have the added benefit of improving the sensitivity of breast cancer screening in young women. Breast density will be employed as a marker of progression-related - proliferative - mechanisms of carcinogenesis.

Secondary study outcomes will include estrogen ratios (catechol estrogen/estradiol), and markers of oxidative DNA damage in peripheral blood and urine (markers of progression-related - mutational - events in carcinogenesis). The responsiveness of these outcomes will suggest the mechanisms through which tamoxifen exerts its preventive effect. Persistence of the markers after one year of treatment may also provide early information about the anticipated duration of the tamoxifen effect.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will include healthy pre-menopausal women, ages 25 to 45 who meet all of the following eligibility criteria:

  * Signed and dated informed consent documents (2) for the study in accordance with all applicable Federal, State and Institutional regulations
  * Lifetime breast cancer risk >20% based on the Gail model, the Claus model, a known familial breast cancer susceptibility mutation, a predicted probability of a BRCA1/2 mutation > 25 % by the Couch model or diagnosis of LCIS or DCIS, or > 20 Gy of external beam radiation delivered to the chest wall.
  * Regular monthly menstrual periods or pre-menopausal defined as cycle occurring every 21 - 35 days
  * Negative serum pregnancy test
  * Prior tubal ligation or willingness to use a non-hormonal barrier method of contraception for two (2) years
  * Prior to randomization, all baseline radiology test results (mammogram, MRI and biopsy, if applicable) must be reviewed to confirm absence of invasive cancer.

Exclusion Criteria:

* Study participants will be excluded if any of the following conditions occur:

  * Absence of or irregular menstrual periods. Irregular menstrual period defined as menstrual cycle occurring < 21 days or > 35 days within the last six months or serum LH > 45.
  * Oral contraceptive or other hormonal treatment within 3 months of study entry. The participant will be considered deferred for 3 months if she agrees to discontinue use of oral contraceptive pills or other hormonal treatment.
  * History or evidence of any malignancy
  * Use of the following concurrent medications: Anticoagulant therapy (e.g. coumarin containing agents and lovanox), estrogens (including Estring), progestins, androgens, or ovarian steroid hormones.
  * Concurrent serious medical illness including:
  * Uncontrolled Diabetes Mellitus (defined as HgA1C > 9.0 %)
  * Uncontrolled hypertension (defined as systolic >180 or diastolic >110 on average of 2 or more readings taken at each of 2 or more visits after initial visit.)
  * Thromboembolic disease (DVT or PE)
  * Cerebrovascular disease (CVA or TIA)
  * Liver disease (AST and/or ALT > 2 X normal)
  * Renal disease (BUN > 30 mg/dl or Creatinine.>2.0 mg/dl)
  * Pregnant or breast feeding
  * Breast implants
  * Prophylactic mastectomy
  * Bilateral oophorectomy (TAH without BSO is permitted)
  * Greater than 3 months of prior participation in a chemoprevention trial or participation in a chemoprevention trial within the last 6 months
  * Prior treatment with tamoxifen for > 3 months duration at any time in the past
  * Prior treatment with Raloxifene for > 3 months duration at any time in the past
  * Contraindications to MRI: presence of implanted metal including pacemaker, ferromagnetic aneurysm clip, other ferromagnetic implant
  * Refusal to undergo MRI

Deferral Criteria:

* Study participants will be deferred from the study for the time period stated if any of the following conditions occur.

  * If a participant has been treated with tamoxifen for less than 3 months, within the last 6 months, she will be deferred for six (6) months from the date of last dose.
  * If a participant has been treated with Raloxifene for less than 3 months, within the last 6 months, she will be deferred for six (6) months from the date of last dose.
  * If a participant is pregnant or breast feeding she will be deferred for six (6) months from the end of pregnancy or breast-feeding. At that time, eligibility status will be re-evaluated.
  * The participant will be considered deferred for three (3) months if she agrees to discontinue use of oral contraceptive pills, has used "emergency contraceptive pill" (ECP or morning after pill) or other hormonal treatment.
  * If the participant has had an open breast biopsy within the last two months or there is a clinical indication for an open breast biopsy, pathology results must be reviewed. If PATHOLOGY is NEGATIVE for invasive cancer, she will be deferred for two (2) months from the date of her last biopsy.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78
Dates: Start 2000-09; Study Completion 2006-07

PRIMARY OUTCOMES:
Breast Density

SECONDARY OUTCOMES:
Biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Susan Domchek, MD, Principal Investigator — University of Pennsylvania
Locations (7):
- United States (6):
  - UCLA Medical Center, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- European Institute of Oncology, Milan, Italy